# Text4Peds: Short Message Service Evaluating Medical Student Education

## Informed Consent

Initial IRB Document Approval Date: 12/8/15

Text4Peds Informed Consent and Recruitment Statement:

Waiver of Written Consent:

- -Implied consent by completing written survey at beginning of the study
- -The research involves minimal risk and involves no procedures for which a written consent is normally required outside of the research context

### SAINT LOUIS UNIVERSITY

Saint Louis University School of Medicine SSM Cardinal Glennon Children's Hospital

# Recruitment Statement for Text4Peds: Medical Student Edition Research Participation

- 1. Christopher Brownsworth, MD, Jamie Sutherell MD, MEd, Associate Professor of Pediatrics, Marta King, MD, MEd, Assistant Professor of Pediatrics, Matthew Schuelke, PhD and Matthew Broom, MD, Assistant Professor of Pediatrics, are inviting you to participate in this research study.
- 2. The purpose of Text4Peds: Medical Student Edition study is to:
  - a. To assess whether texting medical facts to third year medical students in addition to standard educational materials improves performance on the NBME Pediatric Subject Evaluation versus standard educational materials alone
  - b. Assess attitudes towards the Text4Peds program among medical student learners
- 3. Your participation in this study will involve allowing us to use your basic demographic information, program evaluation surveys and your score on the NBME Pediatric Subject Evaluation.
- 4. All study participants will complete a short demographic survey and receive access (through a Google site) to informational material covering common pediatric NBME topics. By completing this baseline survey, you are consenting to participating in the study. Participants will then be randomized to receive a daily question-and-answer (Q&A) text or no text at all. The text message will contain a link to an online site allowing you to answer the question and receive an immediate answer and explanation.
- 5. If you choose not to receive immediate feedback a subsequent text message will be sent, containing the answer to the question. The texts will be sent 6 days/week for 7 weeks for a total of ~42 question and answer texts. At the end of the block, as part of the pediatric clerkship, you will take the NBME Pediatric Subject Evaluation (you will take the test even if you do not participate in the study).
- 6. The risks to you as a participant are minimal. These include breach of confidentiality and receiving incorrect medical knowledge information. To minimize the risk of a breach of confidentiality, the key connecting study ID numbers to names will be stored in a password-protected electronic file on a secure server. All questions, answers and explanations will be reviewed by board certified physicians prior to dissemination of the information. If errors are found after dissemination, the corrected information will be sent by email to you.
- 7. The results of this study may be published in scientific research journals or presented at professional conferences. However, your name and identity will not be revealed and

- your record will remain confidential. Participation will not affect your grade, academic standing, or status.
- 8. Drs. Brownsworth and Broom will have access to all data. Drs. Sutherell, King and Schuelke will have access only to de-identified data. Drs. Sutherell and King would normally have full access to students' NBME data given their responsibilities as course directors for the general pediatrics rotation.
- 9. Participation in this study may benefit you by consistent (2 months) exposure to pediatric medical information which will likely be helpful in the pediatric clerkship and for the pediatric NBME exam. Your participation may benefit others from the determination of whether texting is helpful in adjunct to convey medical information to medical students
- 10. You can choose not to participate. If you decide not to participate, there will not be a penalty to you or loss of any benefits to which you are otherwise entitled. You may withdraw from this study at any time.
- 11. If you have questions about this research study, you can call Christopher Brownsworth, MD at 314-577-5600, or call Matthew Broom, MD at 314-268-4150. If you have questions about your rights as a research participant, you can call the Saint Louis University Institutional Review Board at 314-977-7744 and reference IRB # 26458.



Institutional Review Board 3556 Caroline Street, Room C110 St.Louis, MO 63104

> TEL: 314 977 7744 FAX: 314 977 7730 www.slu.edu

#### NOTICE OF INSTITUTIONAL REVIEW BOARD APPROVAL

Date: December 17, 2015

**To:** Brownsworth, Christopher, Pediatrics

Wilmott, Robert, Pediatrics

From: Kisselev, Oleg, Chairperson, Associate Professor, Minimal Risk #1

Protocol Number: 26458

**Protocol Title:** Text4Peds: Medical Student Edition v. 1

### Sponsor Protocol Version Number and Version Date: Not Applicable

The above-listed protocol was reviewed and approved by the Saint Louis University Institutional Review Board.

Assurance No: FWA00005304

Below are specifics of approval:

Form Type: NEW

Level of Review: EXPEDITED #5, #7

Form Approval Date: December 08, 2015

Protocol Expiry Date: December 07, 2016

HIPAA Compliance: Not Applicable

Waiver of Consent: Waiver of Written Consent

The Saint Louis University Institutional Review Board complies with the regulations outlined in 45 CFR 46, 45 CFR 164, 21 CFR 50 and 21 CFR 56.

Approved Study Documents Include: T1DM Review Article.pdf; Approved\_Text4Peds, Medical Student Edition v1SubjectFlow.pdf; Approved\_Text4PedsExampleQuestion.pdf; Approved\_Text4PedsMedicalStudentEditionv1.0DemographicsSurvey.pdf; Approved\_Text4PedsMedicalStudentEditionv1StudyCompletionEvaluation.pdf; Approved\_Cont.Survey.pdf; Approved\_T4PMedStudentv.1.0RecruitmentStatement.pdf